CLINICAL TRIAL: NCT00589706
Title: A Phase II Study o the Adjuvant Use of Anti-Epidermal Growth Factor Receptor-425 (Anti-EGFR-425) Monoclonal Antibody Radiolabeled With I-125 for High Grade Gliomas
Brief Title: A Phase II Study of Adjuvant Use of Anti-Epidermal Growth Factor Receptor EGFR-425 in High Grade Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12555
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Gliomas
Keywords: high grade gliomas of the brain; anti-body treatment; survival
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A (Experimental): All patients receive the same treatment of MAb-425 +Iodine 125 in a total of three injections. The purpose of this protocol is to allow you to receive course(s) of 1251-MAB 425 until your brain tumor begins to grow, you develop side effects to the treatment, or your medical condition changes (ie: become affected with human immunodeficiency virus (HIV) or develop another cancer).
  Interventions: Drug: MAb-425

INTERVENTIONS:
Drug: MAb-425 — MAb425 anti-epidermal growth receptor) and Iodine-125 will be given as an injection for a total of three treatments each separated by one week.

SUMMARY:
Data from the wistar institute indicated that this anti-body labeled with iodine-125 would localized in the tumor cells of high grade gliomas of the brain. the project combines surgery, radiation therapy, chemotherapy with the labeled antibody in a prospective phase II trial in this disease entity.

DETAILED DESCRIPTION:
This is an open-label Phase II study of postoperative radiation therapy followed by Iodine-125 radiolabeled anti-epidermal-growth-factor-receptor monoclonal antibody (125I-MAB 425) derived from cell cultures for high grade malignant gliomas. Each subject will receive postoperative radiation therapy followed by 6.4 mg of 50 mCi labeled 125I-MAB 425 by injection. This dosing regimen will be given three times generally within a two-week period (days one, eight and 15 of therapy) for a total dose of 19.2 mg of 150 mCi labeled 125I-MAB 425 for each course of therapy. The main objective of this study is to determine if the addition of 125I-MAB 425 to postoperative radiotherapy, with or without change, prolongs absolute survival compared to historical control (postoperative radiation therapy alone) in subjects with histologically proven high grade gliomas. The primary efficacy variable is absolute survival and the secondary target variable will be time to progression of the tumor. Multiple courses will be considered based on the subject's clinical status.

ELIGIBILITY:
Inclusion Criteria:

* all cases above 18 years of age

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1985-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Survival | More than a year
  Potential benefits may include improved long-term survival. All or part of your tumor may be destroyed. You may experience relief of symptoms related to your tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Luther W Brady, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Hahneman Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li L, Quang TS, Gracely EJ, Kim JH, Emrich JG, Yaeger TE, Jenrette JM, Cohen SC, Black P, Brady LW. A Phase II study of anti-epidermal growth factor receptor radioimmunotherapy in the treatment of glioblastoma multiforme. J Neurosurg. 2010 Aug;113(2):192-8. doi: 10.3171/2010.2.JNS091211. PMID 20345222